CLINICAL TRIAL: NCT06546670
Title: A Phase I/II Clinical Study to Investigate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of ITU512 in Healthy Participants and Patients With Sickle Cell Disease
Brief Title: A Phase I/II Study of ITU512 in Healthy Participants and Patients With Sickle Cell Disease
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CITU512A12101; 2024-515696-35-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2024-07-16; First posted 2024-08-09 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Sickle Cell Disease
Keywords: ITU512; Low molecular weight; Small molecule; Sickle cell disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1A (Experimental): Part 1A in healthy participants
  Interventions: Drug: ITU512; Drug: Placebo
- Part 1B (Experimental): Part 1B in healthy participants
  Interventions: Drug: ITU512; Drug: Placebo
- Part 1C (Experimental): Part 1C in healthy participants
  Interventions: Drug: ITU512
- Part 2A (Experimental): Part 2A in patients with sickle cell disease
  Interventions: Drug: ITU512; Drug: Placebo
- Part 2B (Experimental): Part 2B in patients with sickle cell disease
  Interventions: Drug: ITU512; Drug: Placebo
- Part 2C (Experimental): Optional extension in patients with sickle cell disease
  Interventions: Drug: ITU512

INTERVENTIONS:
Drug: ITU512 — ITU512 is an investigational, oral, low molecular weight (LMW) compound.
Drug: Placebo — An inactive substance that looks like and is given the same way as ITU512. The effect(s) of ITU512 will be evaluated against the placebo. Placebos are designed as a control and to have no real effect.
  Arms: Part 1A; Part 1B; Part 2A; Part 2B

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (PK), and preliminary food effect of ITU512 as well as the fetal hemoglobin (HbF)-inducing capacity of ITU512. This will be the first evaluation of the potential therapeutic effect of ITU512 in healthy participants and patients with sickle cell disease (SCD).

DETAILED DESCRIPTION:
This is a global, randomized, Phase I/II study to assess the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary food effect of single-agent ITU512 in adult healthy participants, and safety, tolerability, PK, PD, and efficacy of ITU512 in adolescent and adult patients with sickle cell disease (SCD). The study consists of a first-in-human Phase I study (Part 1) in healthy participants, and a Phase II study (Part 2) in patients with SCD.

Part 1 will comprise of Part 1A, Part 1B, and Part 1C. Part 2 will include Part 2A and 2B and may also include an extension part (Part 2C).

ELIGIBILITY:
Key Inclusion Criteria:

Part 1 (Healthy participants)

* Healthy male participants and female participants of non-childbearing potential between 18-55 years of age
* In good health as determined by the investigator's assessment of medical history, physical examination, vital signs, ECG, and laboratory tests
* Participants must weigh at least 50 kg at screening and first baseline (admission) and must have a body mass index (BMI) within the range of 18.0-32.0 kg/m2 inclusive.

Part 2 (Sickle Cell Disease)

- Male and female participants with a diagnosis of sickle cell disease

Key Exclusion Criteria:

Part 1 (Healthy participants)

* QTcF ≥ 450 msec (as a mean value of triplicates)
* History of arrhythmias
* History of significant illness which has not resolved within two (2) weeks prior to initial dosing
* Women of child-bearing potential (WOCBP)

Part 2 (Sickle Cell Disease)

* Current use of hydroxyurea/hydroxycarbamide (HU/HC)
* QTcF ≥ 450 msec (as a mean value of triplicates)
* History of arrhythmias

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 161 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2029-11-12 (Estimated)

PRIMARY OUTCOMES:
Part 1A, Part 1B, Part 1C: Incidence of AEs and SAEs | Up to approximately 60 days
  Number of participants with adverse events (AEs) and serious adverse events (SAEs), including changes in vital signs, electrocardiograms (ECGs) and laboratory values qualifying and reported as AEs.
Part 1A, Part 1B , Part 1C: Dose discontinued due to AE | Up to 30 days
  Number of participants with dose discontinuation due to AEs
Part 2A, Part 2B: Incidence of AEs and SAEs | Up to 5 months
  Number of participants with adverse events (AEs) and serious adverse events (SAEs), including changes in vital signs, electrocardiograms (ECGs) and laboratory values qualifying and reported as AEs.
Part 2A, Part 2B: Dose interruptions and reductions | Up to 4 months
  Number of participants with dose interruptions or reductions of ITU512
Part 2A, Part 2B: Dose intensity | Up to 4 months
  Dose intensity of ITU512 is computed as the ratio of actual cumulative dose received and actual duration of exposure
Part 2B: Fetal hemoglobin (HbF)% | Month 4
  Assessment of fetal hemoglobin expression by measuring fetal hemoglobin (HbF)% by high-performance liquid chromatography (HPLC) assay

SECONDARY OUTCOMES:
Part 1A, Part 1B: Area under the plasma concentration-time curve (AUC) of ITU512 | From pre-dose up to 144 hours post-dose on Day 1 (Part 1A) and from pre-dose up to 24 hours post-dose on Day 1 and Day 10 (Part 1B)
  Pharmacokinetic (PK) parameters calculated based on ITU512 plasma concentrations by non-compartmental methods
Part 1A, Part 1B: Maximum plasma concentration (Cmax) of ITU512 | From pre-dose up to 144 hours post-dose on Day 1 (Part 1A) and from pre-dose up to 24 hours post-dose on Day 1 and Day 10 (Part 1B)
  PK parameters calculated based on ITU512 plasma concentrations by non-compartmental methods
Part 1A, Part 1B: Time to maximum plasma concentration (Tmax) of ITU512 | From pre-dose up to 144 hours post-dose on Day 1 (Part 1A) and from pre-dose up to 24 hours post-dose on Day 1 and Day 10 (Part 1B)
  PK parameters calculated based on ITU512 plasma concentrations by non-compartmental methods
Part 1A, Part 1B: Renal clearance (CLr) | From pre-dose up to 48 hours post-dose on Day 1 (Part 1A) and from pre-dose up to 24 hours post-dose on Day 1 and Day 10 (Part 1B)
  PK parameters calculated based on ITU512 urine concentrations by non-compartmental methods. The renal clearance (CLr) may be determined based on AUC and amount of drug excreted into urine (Ae) available for the same time period.
Part 2A, Part 2B: Plasma concentrations of ITU512 | From pre-dose up to 4, 6 or 8 hours post-dose on Day 1 at Month 1 and Month 2
  ITU512 concentration in plasma determined in non-placebo treated participants by a validated liquid chromatography with tandem mass spectrometry (LC-MS/MS) method
Part 2A, Part 2B: Urine concentrations of ITU512 | From pre-dose up to 4 or 8 hours post-dose on Day 1 at Month 1
  ITU512 concentration in urine determined in non-placebo treated participants by a LC-MS/MS method
Part 2A: Fetal hemoglobin (HbF)% | Up to 4 months
  Assessment of fetal hemoglobin expression by measuring fetal hemoglobin (HbF)% by HPLC assay
Part 2A, Part 2B: Change from baseline in total hemoglobin (Hb) | Baseline, up to 4 months
  Change from baseline in total hemoglobin (Hb) over time measured in blood samples
Part 1A, Part 1B, Part 2A, Part 2B: Change from baseline in Fridericia- corrected Holter QT interval (QTcF) | Up to 4 months
  Real-time 12-lead safety ECGs will be locally collected and evaluated. Change from baseline in QTcF with respect to PK parameters and/or ITU512 concentrations will be assessed
Part 1C: Area under the plasma concentration-time curve from time 0 up to the time of the last quantifiable concentration (AUClast) of ITU512 | From pre-dose up to 144 hours post-dose
  PK parameters calculated based on ITU512 plasma concentrations by non-compartmental methods
Part 1C: Area under the plasma concentration-time curve from time 0 up to infinity (AUCinf) of ITU512 | From pre-dose up to 144 hours post-dose
  PK parameters calculated based on ITU512 plasma concentrations by non-compartmental methods
Part 1C: Maximum plasma concentration (Cmax) of ITU512 | From pre-dose up to 144 hours post-dose
  PK parameters calculated based on ITU512 plasma concentrations by non-compartmental methods
Part 1C: Time to maximum plasma concentration (Tmax) of ITU512 | From pre-dose up to 144 hours post-dose
  PK parameters calculated based on ITU512 plasma concentrations by non-compartmental methods

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Sciences Sea View, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.